CLINICAL TRIAL: NCT05352646
Title: Autologous Memory Lymphocyte（NewishT）for Hepatocellular Carcinoma With High Risk of Recurrence After Radical Resection
Brief Title: NewishT Cell Therapy for HCC With High Risk of Recurrence After Radical Resection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newish Technology (Beijing) Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NewishT-HCC-002
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NewishT (Experimental): This study is divided into two dose groups and two phases. Phase Ia climbed from low-dose group to high-dose group in turn according to the 3+3 dose escalation principle. Phase Ib extended 10 subjects each group.
  Interventions: Drug: Autologous memory lymphocyte Injection (NewishT), low-dose group; Drug: Autologous memory lymphocyte Injection (NewishT), high-dose group

INTERVENTIONS:
Drug: Autologous memory lymphocyte Injection (NewishT), low-dose group — Recruited participants in low-dose group will receive autologous memory lymphocyte (NewishT) intravenous infusion every 4 weeks, a total of 2 times.
  Other Names: Low-dose group
Drug: Autologous memory lymphocyte Injection (NewishT), high-dose group — Recruited participants in high-dose group will receive autologous memory lymphocyte (NewishT) intravenous infusion every 2 weeks, a total of 4 times.
  Other Names: High-dose group

SUMMARY:
This is a single-arm, open label, multi-center Phase 1 clinical study to evaluate the safety and efficacy of autologous memory lymphocyte therapy (NewishT) in patients with hepatocellular carcinoma at high risk of recurrence after radical resection.

DETAILED DESCRIPTION:
This study is divided into two dose groups and two phases. Phase Ia climbed from low-dose group to high-dose group in turn according to the 3+3 dose escalation principle. Phase Ib extended 10 subjects each group.

After the completion of treatment, the subjects shall continue to receive safety follow-up until 14 days after the last administration, and all adverse events shall revert to level I or all adverse events shall be clinically stable (whichever is later achieved); Tumor imaging assessment was performed at week 7 and week 20 to observe the progression of disease.

After week 20, the survival follow-up period was entered, and patients were followed up until death, loss of follow-up, or trial termination, whichever occurred first. Survival was followed up by telephone every 12 weeks (±7 days), and radiographic evidence should be obtained if recurrence/progression occurred.

ELIGIBILITY:
Inclusion criteria:

Patients had to meet all of the following inclusion criteria:

1. 18≤ age ≤75, regardless of gender;
2. Primary hepatocellular carcinoma, which was diagnosed in one of the following conditions: 1) Hepatocellular carcinoma (HCC) confirmed by histopathology or cytology; 2) Meet the clinical diagnostic criteria of liver cancer in the Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2022 edition);
3. HBsAg or HBV DNA positive serological test, active virus infection is willing to accept anti-HBV virus treatment during the study period;
4. Barcelona clinic liver cancer (BCLC) stage A/B or Chinese Hepatocellular carcinoma Stage (CNLC) IA-IIIA;
5. Underwent radical resection of liver cancer (open surgery, laparoscopic surgery, ablation, robot-assisted surgery) within 12 weeks before blood sampling for the first NewishT preparation; The interval between clinical staging of BCLC or CNLC hepatocellular carcinoma and radical resection was less than 12 weeks.
6. No residual intrahepatic tumor was found by imaging examination within 4 weeks before blood sampling for the first NewishT preparation; No lymph node metastasis, no extrahepatic metastasis;
7. Patients undergoing radical resection of liver cancer should meet the intraoperative criteria of radical resection of liver cancer:

(1) There was no invasion of adjacent organs, hilar lymph nodes or distant metastasis during the operation; (2) Negative cutting margin;

8. No Vp4 macrovascular invasion, hepatic vein or inferior vena cava macrovascular invasion of any grade after radical resection (see Appendix 12 for definition of macrovascular invasion);

9. Meeting any of the following high recurrence risk factors after radical mastectomy:

Patients undergoing radical resection:

1. Number of tumors ≥3;
2. Single tumor patients: patients with tumor diameter ≥ 5cm;
3. Single tumor patients: patients with tumor diameter < 5cm, pathological report showed Microvascular invasion (MVI) or Vp1/Vp2/Vp3 macrovascular invasion;
4. Edmondson-Steiner grade Ⅲ or Ⅳ of hepatocellular carcinoma;

Patients undergoing radical ablation:

1. Patients with multiple tumors: the diameter of all tumors ≤5cm and the number of tumors ≤4;
2. Single tumor patients: tumor diameter 2-5cm;
3. Edmondson-Steiner grade Ⅲ or Ⅳ of hepatocellular carcinoma ;

10. Within 1 week before blood collection for the first NewishT preparation, ECOG performance status score was 0-1;

11. Child-Pugh score A/B (≤7) within 1 week before blood collection for the first NewishT preparation;

12. Major organ functions were normal within 1 week before blood collection for the first NewishT preparation:

Blood routine:

Hemoglobin (Hb) ≥75 g/L (no infusion of concentrated red blood cells or erythropoietin within 2 weeks); Absolute neutrophil count (ANC) ≥1.5×109/L (no granulocyte colony-stimulating factor was used within 2 weeks); Absolute lymphocyte count (LYMP) ≥0.8×109/L; (4) Platelet count (PLT) ≥50×109/L;

The liver:

Total bilirubin (TB) ≤3× upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN; Plasma albumin ≥28g/L;

Blood coagulation function:

International normalized ratio (INR) ≤2.3;

Kidney:

Serum creatinine (Scr) ≤1.5×ULN, or creatinine clearance ≥50 mL/min (serum creatinine > 1.5 x ULN);

13. The expected survival time is more than 6 months;

14. Within 1 week before blood collection for the first NewishT preparation, women of childbearing age must have a negative serum pregnancy test and consent to use effective contraception during the use of the study drug and within 6 months after the last administration of the study drug. For men, they should be surgically sterilized or agree to use effective contraception during study drug use and for 6 months after the last administration of study drug.

15. Have fully understood the study and voluntarily signed the ICF, have good communication with the investigator, and are able to complete all treatments, examinations, and visits stipulated in the study protocol.

Exclusion criteria:

Patients with any of the following were excluded from the study:

1. HCC recurred before blood collection for the first NewishT preparation;
2. Before blood sampling for the first NewishT preparation, the investigator judged that the patient had not fully recovered from the toxicity and/or complications of radical resection;
3. There are contraindications to TACE;
4. After radical hepatectomy or during the screening period, received or planned to receive radiotherapy, chemotherapy, molecular targeted therapy, biological therapy, TACE therapy, radiofrequency ablation and other anti-liver cancer therapies (except postoperative TACE adjuvant therapy specified in the protocol);
5. accompanied by hepatic encephalopathy;
6. Regular renal dialysis is required;
7. with uncontrolled pleural effusion, pericardial effusion, or moderate or more ascites (refers to ascites that cannot be easily controlled by diuretic treatment);
8. A history of gastrointestinal bleeding, current active bleeding, or bleeding tendency within 28 days before screening;
9. had received systemic antitumor therapy (including chemotherapy, molecular targeted therapy, biological immunotherapy) for liver cancer within 28 days before screening;
10. had undergone transcatheter arterial interventional therapy (transcatheter arterial chemoembolization [TACE], transcatheter arterial chemoembolization [TAE], transcatheter arterial infusion chemotherapy [HAIC], radioactive microsphere TACE[TARE], etc.), radiotherapy, microwave ablation, cryotherapy, high-power ultrasound focused ablation and other local treatments for liver tumors. Radical ablation and resection are excluded;
11. Participated in another clinical trial or was under observation in another clinical trial within 28 days prior to screening;
12. Continuous (more than 1 week) glucocorticoid therapy (dose equivalent to prednisone > 10 mg/ day), except hormone replacement therapy and intratracheal administration;
13. A history of immune deficiency or autoimmune diseases (e.g., rheumatoid joint disease, systemic lupus erythematosus, multiple sclerosis, etc.);
14. A history of allogeneic stem cell/tissue/solid organ transplantation (including bone marrow transplantation);
15. with uncontrolled severe infection (> grade 2 NCI-CTC adverse events, version 5.0);
16. Persons with a history of hepatitis C virus (HCV) infection or human immunodeficiency virus (HIV) infection or carriers of syphilis;
17. Patients with serious other organ dysfunction or cardiopulmonary diseases;
18. epilepsy that requires treatment with medication (e.g. steroids or antiepileptic drugs);
19. had or currently has other malignancies (with the exception of adequately treated and completely cured ductal carcinoma in situ of the breast, carcinoma in situ of the cervix, basal cell carcinoma of the skin, superficial bladder tumor, or any malignancy that was cured more than 5 years before study entry);
20. a known history of albumin allergy, or severe allergy, or allergic disease, or allergic constitution, or severe iodine contrast allergy, meeting any of these criteria;
21. severe mental illness;
22. a history of drug or alcohol abuse;
23. pregnant or lactating women, or women of childbearing age with positive blood pregnancy tests, or patients of childbearing age and their spouses are unwilling to use effective contraception during and within 6 months after the completion of the clinical study;
24. Patients deemed by the investigator to be ineligible for this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity (DLT) | 14 days after last administration
  Any AEs that is definitely, probably, or possibly related to the test drug occurring within 14 days of the last dosing will be classified as DLT during dosing climb.

SECONDARY OUTCOMES:
All adverse events (AE) | 1 year
  Including incidence and severity of serious adverse events (SAE) (according to NCI-CTCAE Standard version 5.0 of common Terms for Adverse Events)
recurrence-free survival(RFS) rate | 1 year
  The probability of no recurrence or death within 1 year from the date of radical hepatocellular carcinoma resection.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiang Cai, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: by publication